CLINICAL TRIAL: NCT03697577
Title: Pilot Study Assessing the Effect of Cyclin-dependent Kinase 4/6 Inhibitors on Body Composition in Patients With ER+/HER2- Metastatic Breast Cancer
Brief Title: CDK and Body Composition Study
Status: Recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-9567
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: cyclin-dependent kinase (CDK) 4/6 inhibitors; Body composition; body fat mass; metastatic ER+/HER2- breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tomography, X-Ray Computed; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Total Number of Specimens 60 Project/Storage Duration: 24 Months Sample Type: BLOOD-SERUM Specimen Volume: 15cubic centimeters (15cc) Sample Preservation Measures: STANDARD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ER+/HER2- metastatic breast cancer: Subjects have metastatic ER+/HER2- breast cancer, and their doctor is offering treatment with CDK 4/6 inhibitors as standard of care treatment. It is hypothesized that cyclin-dependent kinase (CDK) 4/6 inhibitors decrease fat mass among women with ER+/HER2- metastatic breast cancer without significant effect in the skeletal mass. Body composition will be obtained from CT scans (CT or PETCT) as part of standard of care, and body fat mass will be obtained from DEXA scan (DEXA will be performed only if available)
  Interventions: Diagnostic Test: CT scans; Diagnostic Test: DEXA scan

INTERVENTIONS:
Diagnostic Test: CT scans — Patients will undergo CT or PETCT as part of standard of care
Diagnostic Test: DEXA scan — Patients will undergo DEXA scan to measure body fat mass (DEXA will be performed only if available)

SUMMARY:
The goal of this study is to evaluate changes in body composition among patients who are treated with cyclin-dependent kinase (CDK) 4/6 inhibitors (abemaciclib, ribociclib, or palbociclib).

DETAILED DESCRIPTION:
The goal of this study is to evaluate changes in body composition among patients who are treated with cyclin-dependent kinase (CDK) 4/6 inhibitors (abemaciclib, ribociclib, or palbociclib). There is preliminary data suggesting that these drugs have more effect on body fat mass than body muscle mass. These drugs have already been approved by U.S Food and Drug Administration (FDA) to treat ER+/HER2- metastatic breast cancer. The investigators will follow up body composition changes among patients who receive CDK 4/6 inhibitors as part of their standard of care. Body composition changes will be measured from Computed Tomography (CT) or Positron Emission Tomography/Computed Tomography (PET/CT) scans that are part of standard of care treatment, and from DEXA scans (DEXA is optional and will be performed only if available). The investigators will also conduct body measurements with measuring tape and will draw blood tests to assess for fat biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast that is Estrogen Receptor (ER) and/or Progesterone Receptor (PR) positive based on current American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) guidelines
* Metastatic or locally advanced/inflammatory, unresectable breast cancer not amenable to potentially curative surgery
* Measurable and/or non-measurable as defined by RECIST 1.1 criteria
* Patients must be a candidate to start an FDA approved CDK 4/6 inhibitor (palbociclib, ribociclib, abemaciclib) as part of standard of care treatment
* Female, or male patients, and age >=18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Ability to understand and the willingness to sign a written informed consent document
* Concomitant therapy with bisphosphonates, RANKL inhibitors or growth-colony-stimulating factor (G-CSF) is allowed as per physician decision

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CDK 4/6 inhibitors or other agents used in the study (e.g., fulvestrant, letrozole, anastrozole, exemestane)
* BMI < 18.5
* Prior CDK 4/6 use in any setting
* Inability to undergo anthropometric measurements
* Inability to undergo CT scan imaging
* Women of child-bearing potential must not be pregnant or breast feeding. They must also agree to use adequate contraception (hormonal or barrier method of birth control) and not be breast feeding prior to study entry, for the duration of study participation, and for up to 10 days after completion of all protocol therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study or up to 10 days after completion of protocol therapy, she should inform her treating physician immediately
* Intercurrent illness that would substantially increase the risk of treatment associated complications (e.g., active infection, uncontrolled diabetes mellitus or hypertension)
* Psychiatric illness/social situations that would interfere with the patient's ability to comply with the treatment regimen
* Patients with untreated brain metastasis are excluded. Patients with a prior history of brain metastasis are eligible if they have received prior brain radiation (whole brain or stereotactic radiosurgery) or surgery, have stable intracranial disease for at least 3 months after completion of local therapy, and are not taking corticosteroids for treatment of brain metastasis
* Patients who have not recovered (i.e., CTCAE Grade ≤1 or baseline) from an adverse event due to a previously administered agent, excluding alopecia
* Patients with inability to swallow and retain pills
* Malabsorption syndrome or other gastrointestinal illness that could affect oral absorption
* Patients with active implanted medical devices (cardiac pacemakers, defibrillators or patients connected to electronic life support devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being asked to participate in this study because they have metastatic ER+/HER2- breast cancer, and their doctor is offering treatment with CDK 4/6 inhibitors as standard of care treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Total adipose tissue (TAT) | From Baseline and 6 months after CDK 4/6 inhibitor therapy
  Total Adipose tissue (TAT) is defined as the sum of intramuscular adipose tissue (IMAT), visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT) obtained from L3 cross section from CT scans. Only patients who complete 24 weeks of CDK 4/6 inhibitor treatment and have no radiological/clinical signs of disease progression will be included in the analysis of primary endpoint. Results will be calculated and summarized in area (cm²).

SECONDARY OUTCOMES:
Body Fat Mass (BFM) using Dual-energy X-ray Absorptiometry (DEXA) | Baseline and 6 months after CDK 4/6 inhibitor therapy
  Body Fat Mass will be obtained from dual-energy x-ray absorptiometry (DEXA). The DEXA scan calculates the ratio of soft tissue attenuation at different X-ray energies. Results are measured and reported in kilograms (kg). DEXA scans are optional and will be performed only if available.
Body Lean Mass (BLM) using Dual-energy X-ray Absorptiometry (DEXA) | Baseline and 6 months after CDK 4/6 inhibitor therapy
  Body Lean Mass (BLM) will be obtained from dual-energy x-ray absorptiometry (DEXA). The DEXA scan calculates the ratio of soft tissue attenuation at different X-ray energies. Results are measured and reported in kilograms (kg). DEXA scans are optional and will be performed only if available.
Skeletal muscle index (SMI) | Baseline and 6 months after CDK 4/6 inhibitor therapy
  Skeletal muscle index (SMI) will be obtained by dual-energy x-ray absorptiometry (DEXA). The DEXA scan will be used to measure the amount of lean muscle in the body. SMI is defined as muscle area at L3 cross section from CT scans in cm^2 divided by height in meters squared. DEXA scans are optional and will be performed only if available.
Adipose Serum Biomarkers - Fasting Glucose | Baseline and 3 months and 6 months after CDK 4/6 inhibitor therapy
  Fasting glucose levels in blood sera will be measured using a glucose blood sugar test. Normal ranges vary based on the health of the individual however standard glucose concentrations are between 70 mg/dL (3.9 mmol/L) -100 mg/dL (5.6 mmol/L). Glucose levels between 100-125 mg/dL (5.6-6.9 mmol/L) may be indicative of prediabetes. Fasting glucose levels >126 mg/dL on successive tests is correlated with diabetes. Results will be summarized and reported.
Adipose Serum Biomarkers - Lipid Panel (Total Cholesterol and LDL cholesterol, HDL cholesterol, and Triglycerides) | Baseline and 3 months and 6 months after CDK 4/6 inhibitor therapy
  A lipid panel will be used to assess Total cholesterol, LDL Cholesterol, HDL Cholesterol, and triglyceride levels in blood sera samples. Each parameter has unique ranges and can vary by age, weight, and sex; however, High concentrations of Total cholesterol and LDL cholesterol increases the risk of coronary heart disease and atherosclerosis. HDL cholesterol ("good cholesterol") removes excess cholesterol from the body. High triglyceride levels also increase the risk of cardiovascular disease. Results for each parameter will be summarized and reported in mg/dL.
Adipose Serum Biomarkers - Dehydroepiandrosterone Sulphate (DHEAS) | Baseline and 3 months and 6 months after CDK 4/6 therapy
  DHEAS levels in blood sera will be measured using a DHEA-sulfate (DHEAS) blood test. This test can be used to check the function of the adrenal glands. Normal ranges vary based on age, gender and laboratory; however, high concentrations could be indicative of adrenal tumors, Cushing's disease, polycystic ovary syndrome (PCOS), or adrenal hyperplasia. Results will be summarized and reported in ug/dL.
Adipose Serum Biomarkers - Insulin | Baseline and 3 months and 6 months after CDK 4/6 inhibitor therapy
  Insulin levels in blood sera will be measured using an insulin blood test. Insulin is a hormone that regulates glucose absorption. Normal ranges vary based on the type of test administered and the health of the individual; however, standard fasting insulin concentrations are usually <25 mIU/L. Higher concentrations can be indicative of insulin resistance. Results will be summarized and reported.
Adipose Serum Biomarkers - Leptin | Baseline and 3 months and 6 months after CDK 4/6 inhibitor therapy
  Leptin will be assessed using a leptin blood test that measures the concentration of leptin in blood sera. Leptin is a hormone that helps regulate appetite and energy levels. Standard ranges vary based on age, gender, body mass index, and other variables; however, ranges are generally between 0.5-15.2 ng/mL for females and 0.5-12.5 ng/mL for males. Results will be summarized and reported.
Adipose Serum Biomarkers - Free Leptin Index (FLI) | Baseline and 3 months and 6 months after CDK 4/6 inhibitor therapy
  FLI will be assessed by blood test and calculated as the ratio of total leptin and soluble leptin receptor (sOB-R) concentrations. FLI is a biomarker of leptin resistance and the status of leptin action. High FLI is a risk factor for obesity and is associated with several chronic diseases. Results will be summarized and reported.
Adipose Serum Biomarkers - Adiponectin | Baseline and 3 months and 6 months after CDK 4/6 inhibitor therapy
  Adiponectin will be assessed using an adiponectin test that measures the concentration of adiponectin in the blood. Adiponectin is a protein hormone produced by fat cells that helps regulate blood sugar and fat metabolism. Lower levels of adiponectin in blood sera are often linked to conditions like obesity, type 2 diabetes, and heart disease. A normal adiponectin blood test result is generally 5-30 ug/mL but can vary depending on age and body mass index (BMI). Results will be summarized and reported.
Adipose Serum Biomarkers - High-sensitivity C-reactive protein (hsCRP) | Baseline and 3 months and 6 months after CDK 4/6 inhibitor therapy
  hsCRP will be measured and reported by blood test. hsCRP measures the concentration of C-reactive protein (CRP) in blood. CRP is a protein that increases in response to inflammation and is correlated with adverse cardiovascular and cerebrovascular outcomes. Normal results are generally risk stratified with concentrations <1.0 mg/dL indicating a low risk of cardiovascular disease; concentrations between 1.0-3.0 mg/dL indicating an average risk of cardiovascular disease; and concentrations >3.0 mg/dL indicating a high risk of cardiovascular disease. Results will be summarized and reported.
Body Fat Mass (BFM) using Bioimpedance spectroscopy (BIS) | Baseline and 3 months and 6 months after CDK 4/6 inhibitor therapy, and every 3 months thereafter up to 24 months
  BFM will be measured with the use of bioimpedance spectroscopy (BIS). BIS is a non-invasive method that takes measurements at 256 different frequencies and uses mathematical modeling to calculate electrical resistance throughout the body. Fat tissue has significantly higher resistance compared to lean muscle tissue. The total weight of body fat estimated by the BIS analysis will be expressed in kilograms and summarized for the group.
Body Fat-Free Mass (FFM) | Baseline and 3 months and 6 months after CDK 4/6 inhibitor therapy, and every 3 months thereafter up to 24 months
  FFM will be derived based on the BFM readout obtained from the BIS analysis. The "fat-free mass" will be calculated by subtracting the total body weight minus the estimated BFM obtained by BIS analysis, based on electrical resistance through the body. This result will be expressed in kilograms and summarized for the group.
Anthropometric measurements - Body Mass Index (BMI) | Baseline and every 4 weeks for the first 6 months after CDK 4/6 inhibitor therapy and every 3 months thereafter up to 24 months
  BMI will be determined by obtaining height and body weight measurements. It is calculated by dividing body weight in kilograms (kg) by height in meters squared (m^2). A BMI of 30 kg/m^2 or higher has been used to define obesity in most reports, including those showing an association between obesity and increased risk of cancers, cancer mortality, and mortality from all causes. Group results will be summarized and reported.
Anthropometric measurements - Skin fold thickness (biceps, triceps, subscapular, and suprailiac) | Baseline and every 4 weeks for the first 6 months after CDK 4/6 inhibitor therapy and every 3 months thereafter up to 24 months
  Skin fold thickness will be measured with the use of calipers. Skin fold thickness measurements will be obtained for the biceps, triceps, subscapular, and suprailiac sites. Calipers will be used to pinch the skin and lift it away from the muscle at each site and measure the thickness of skin folds at each location. Values will be summarized in millimeters (mm) for the group and reported. Skin fold thickness measurements provide an overall picture of subcutaneous fat distribution.
Anthropometric measurements - Abdominal circumference | Baseline and every 4 weeks for the first 6 months after CDK 4/6 inhibitor therapy and every 3 months thereafter up to 24 months
  Abdominal circumference is a measurement of the horizontal distance around the abdomen. Abdominal circumference will be assessed by determining the midpoint between the lower rib margin and the iliac crest and measuring the circumference at the midpoint, in centimeters, with measuring tape while breathing normally. Group results will be summarized. An enlarged abdominal circumference can be a sign of obesity and a risk factor for disease.
Anthropometric measurements - Waist-to-hip ratio | Baseline and every 4 weeks for the first 6 months after CDK 4/6 inhibitor therapy and every 3 months thereafter up to 24 months
  Waist-to-hip ratio will be measured with measuring tape by measuring the narrowest part of the waist followed by the widest part of the hips and dividing the waist measurement by the hip measurement. While normal values can vary, a healthy waist-to-hip ratio is generally considered to be below 0.9 for men and 0.85 for women, according to the World Health Organization (WHO). Group results will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Anampa, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No